CLINICAL TRIAL: NCT05772364
Title: Metabolic Response to the Consumption of Waters With Different Calcium Content: a Cross-over Clinical Study
Brief Title: High- Versus Low-calcium Water for Bone Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CALIMOS (PI: M Briguglio); L4179 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Orthopedic Disorder; Calcium Metabolism Disorders; Bone Resorption; Water-Electrolyte Imbalance; Eating, Healthy
MeSH Terms: conditions — Musculoskeletal Diseases; Calcium Metabolism Disorders; Bone Resorption; Water-Electrolyte Imbalance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-calcium water first, then high-calcium water (Experimental): Participants drink 1.5 L of the designated water
  Interventions: Other: Loading of low-calcium water first, then high-calcium water

INTERVENTIONS:
Other: Loading of low-calcium water first, then high-calcium water — All cohort subjects are asked to consume water with less than 5 mg/L of calcium first, then are asked to consume water with at least 400 mg/L of calcium

SUMMARY:
The experimental study investigates which metabolic responses of calcium and parathyroid hormone are observable in blood and urine in a cohort of 41 healthy adults following a sequence of different exposures: low-calcium water first and high-calcium water afterward.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 18 and < 30
* Maintenance of diet and physical activity lifestyle throughout the duration of the study
* Acceptance of informed consent

Exclusion Criteria:

* Consumption of water with calcium > 150 mg/L
* Pregnancy (as established by self-declaration), breastfeeding, menopause
* Inability to follow the study protocol
* Cardiac, vascular, renal, and oncological disease
* Neuropsychiatric disease, developmental disorders
* Disease or past surgery affecting the gastrointestinal tract
* Drugs that interfere with bone (e.g. corticosteroids) or with fluid balance (e.g. diuretics)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change of blood calcium levels | Baseline and 2.5 hours
  Change of calcium levels (mg/dL) from baseline and after 2.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Briguglio, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided